CLINICAL TRIAL: NCT04379791
Title: Factors Influencing the Risk of Surgical Site Infections and Wound Complications in Operatively Treated Ankle Fractures in the Elderly - a Case Control Study
Brief Title: Factors Influencing the Risk of Surgical Site Infections and Wound Complications in Operatively Treated Ankle Fractures in the Elderly
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00318; ch20Eckardt
Record Dates: First submitted 2020-05-06; First posted 2020-05-07 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Ankle Fractures
Keywords: surgical site infections; wound complications; operatively treated ankle fractures; delayed wound healing
MeSH Terms: conditions — Ankle Fractures; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case cohort: Patients with a surgical site infection or a wound complication after surgical treatment of an ankle fracture. The time horizon for wound complication was set to maximally 4 weeks after surgery.
  Interventions: Other: Data collection from routine medical records
- control cohort: Patients without a surgical site infection or a wound complication (normal wound-healing and suture or staple removal) after surgical treatment of an ankle fracture.
  Interventions: Other: Data collection from routine medical records

INTERVENTIONS:
Other: Data collection from routine medical records — Data collection from routine medical records for criteria for fracture related infections (FRI) and for wound complications. Data collection from routine medical records for risk factors.

SUMMARY:
This study is to analyse risk factors for wound complications or surgical site infections and to analyse whether risk factors for wound complications or surgical site infections are also factors for other complications. Based on the data from this study it will be investigated whether a risk score can be build up to predict individual risk for a complication after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 50 years with ankle fractures surgically treated at the University Hospital Basel
* Sufficient Follow up at the University Hospital Basel in order to judge wound healing complications over a 4 weeks period and fracture related infection over a 3 months period

Exclusion Criteria:

* Existence of a documented dissent.
* Distal tibia fractures and Pilon fractures
* Followed up at another institution or with no follow up at our institution for any other reason

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ankle fractures surgically treated at the University Hospital Basel starting with the patients operated in 2017 and then going backwards in time, until 120 patients with a surgical site infection or a wound complication are found. Then randomly collection of 120 controls among the remaining investigated patients .
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
association between single risk factors and outcome (wound healing complication, surgical site infection) | at Baseline
  In a first step analyses of the association between single risk factors and outcomes will be made. Odds ratios will be reported together with confidence intervals and p-values. In a second step it will be analyzed whether risk factors can be combined into a risk score using Tibshirani's Lasso.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Eckardt, PD Dr. med., Principal Investigator — Dep. of Orthopedics and Traumatology, University Hospital Basel
Locations (1):
- Dep. of Orthopedics and Traumatology, University Hospital Basel, Basel, Switzerland